OFFICIAL USE ONLY
Doc Name : Informed Consent Form Template
Doc Number : 207-001
Doc Version : 13
Date : 31 Jan 2022

#### PARTICIPANT INFORMATION SHEET AND CONSENT FORM

You / Your child are invited to participate in a research study. Please read the information provided, it is important that you / your child understand the information provided in this sheet. You / Your child are welcome to ask any questions before your child consents to participate in this study. If you / your child have any questions on this research study, please see the sections below for our contact information. Should you/ your child agree to participate in this study, please complete the online consent form together with your parent/ child.

# 1. Study Information

#### **Protocol Title:**

Integrative Adolescence Research Programme (IARP) – iAdoRe study

## **Principal Investigator & Contact Details:**

Professor Johan Eriksson Singapore Institute for Clinical Sciences (SICS) Brenner Center, 30 Medical Drive, Singapore 117609 Email: Johan\_eriksson@sics.a-star.edu.sg

Tel: 8854 6302

## 2. Purpose of the Research Study

The purpose of this study is to deepen our understanding of health and well-being, focusing on maximising potential of adolescents in Singapore. The research study is done in collaboration between A\*STAR Singapore Institute for Clinical Sciences (SICS) and National Institute of Education (NIE). You / Your child are invited to participate in this study because you/ your child are enrolled in the *DREAMS* (*Drivers, Enablers and pathways of Adolescent development in Singapore*) cohort study. This study targets to recruit about 1000 - 1200 adolescents, aged 13 – 15 years old, from the *DREAMS* cohort study over a period of 12 months.

#### 3. What procedures will be followed in this study

## Online questionnaires

If you /your child agree to take part in this study, you/ your child will be invited to complete a series of online questionnaires at 2 time points over 2 years, to help us better understand your / your child's health, socio-behavioral development and well-being. The set of online questionnaires for each timepoint will be completed in 2 rounds (according to time availability) and total time taken is estimated to be 2 hours.

Any individually-identifiable data obtained during the course of this study will be stored and analysed for the purposes of this study and future related studies. There are no biological samples collected from this study.

The online questionnaires used in this study are for epidemiological use and not for diagnostic/ medical purposes. However, during the course of the study, there is a possibility that we might unintentionally come to know of new information about you /your child's mental well-being from the questionnaires completed in the study. These are called "incidental findings".

"Incidental findings" are findings that have potential health importance to research participants like you/ your child and are discovered in the course of conducting the study, but are unrelated to the purposes, objectives or variables of the study.

If any potential incidental findings regarding profile of mental health concerns (e.g., eating problems, depressive symptoms or bullying) and/or risk of serious harm are identified during the course of this study, we will inform the school counsellor to ensure the safety and well-being of you / your child. The school counsellor will then notify you / your child and may conduct further evaluations as needed.

It is important to note that while we may bring such results to the school counsellor, we want to make it clear that you / your child should not rely on this study for information on the state of your / your child's health for your / your child medical care and management. We kindly advise you / your child to consult a healthcare professional for further investigation.

The costs for any care that will be needed to diagnose or treat any incidental finding would not be paid for by this research study. These costs would be your / your child responsibility.

# 4. Your Responsibilities in This Study

Should you / your child agree to participate in this study, you / your child will complete a series of online questionnaires at 2 timepoints. You / your child may choose to end the participation in this study at any time.

## 5. What Is Not Standard Care or is Experimental in This Study

This study participation is not part of your / your child's clinical care and are only meant for research purposes. All data collected concerning you / your child will be used strictly for research purposes only.

#### 6. Possible Risks and Side Effects

There are no risks to individuals participating in this study. We anticipate little or no discomforts involved when completing the questionnaires. There will be minimal disruption to your / your child's school's curriculum.

There may be some questions related to sensitive topics (e.g. mental health and puberty). You / your child may choose to skip the questions if you / your child feel uncomfortable. If your / your child's responses show signs of distress, helplines numbers will be shared with you / your child at the end of the questionnaire. Also, study team will inform your / your child's school counsellor to follow-up.

There is a minimal risk of breach of privacy and confidentiality in the study. All personal identifiers (e.g. name, email address) and data collected from this study will be securely stored and protected. Identifiable personal data will only be accessible by delegated study team members.

## 7. Possible Benefits from Participating in the Study

We seek your / your child's understanding that there is no direct benefit from participating in this study. However, your / your child's participation is highly valued and appreciated as it contributes to advancing our knowledge of adolescent health and well-being in Singapore.

## 8. Costs & Payments if Participating in the Study

There are no costs involved if you / your child take part in the study. You / Your child will be reimbursed for your / his / her time and effort. Upon successful completion of all questionnaires at each timepoint, you / your child will receive \$50 worth of gift vouchers. You / your child will receive a total of \$100 worth of gift vouchers for your / his / her participation.

# 9. Voluntary Participation and Compensation for Injury

Your / your child's participation in this study is entirely voluntary, and you/ your child have the right to withdraw from the study at any time without any penalty.

If you / your child decides to stop taking part in this study, you / your child should inform the study team via email / phone. However, the data that has been collected until the time of your / your child's withdrawal will be kept and analysed. The reason is to enable a complete and comprehensive evaluation of the study.

In the event of any new information becoming available that may be relevant to your / your child willingness to continue in this study, you / your child will be informed in a timely manner by the Principal Investigator or his / her representative and further consent may be required.

While no injuries are anticipated in this study, SICS without legal commitment will compensate you / your child for the injuries arising from your / your child's participation in the study without you / your child having to prove SICS is at fault. There are however conditions and limitations to the extent of compensation provided. You / Your child may wish to discuss this with the Principal Investigator.

By agreeing to participate in the study, you / your child will not waive any of your / your child's legal rights or release the parties involved in this study from liability for negligence.

# 10. Confidentiality of Study and Medical Records

Your / your child's participation in this study will involve the collection of "Personal Data". "Personal Data" means data about you / your child which makes you / your child identifiable (i) from such data, or (ii) from that data and other information which an organisation has or likely to have access. Examples of personal data can include your name, nationality, date of birth and telephone number.

Information and "Personal Data" collected for this study will be kept confidential. Your / your child's records, to the extent of the applicable laws and regulations, will not be made publicly available.

To protect your / your child's confidentiality, research data collected will be coded and identifying information will be removed. Your / your child's personal data will never be used in publications, presentations, or future research. The link between you / your child's own identifiable information and the code number will be locked and may only be accessed by the study team and trusted third parties.

However, the Regulatory Agencies, Institutional Review Board and auditors will be granted direct access to your / your child's study records to verify study procedures and data, without making any of your / your child's information public.

Research arising in the future, based on your / your's child "Personal Data" will be subject to review by the relevant institutional review board.

#### 11. Who To Contact if You Have Questions

If you/ your child have questions about this research study, please contact the Principal Investigator or research team at <a href="mailto:idealcolor: blue contact the principal law study co

The study has been reviewed by the NHG Domain Specific Review Board (the central ethics committee) for ethics approval.

If you/ your child want an independent opinion to discuss problems and questions, obtain information and offer inputs on your / your child's rights as a research subject, you / your child may contact the NHG Domain Specific Review Board Secretariat at 6471-3266. You / your child can also find more information about participating in clinical research, the NHG Domain Specific Review Board and its review processes at <a href="www.research.nhg.com.sg">www.research.nhg.com.sg</a>.

If you/ your child have any complaints or feedback about this research study, you/ your child may contact the Principal Investigator or the NHG Domain Specific Review Board Secretariat.